CLINICAL TRIAL: NCT06325358
Title: EXPOSITION (EXPosome, Oxidative Stress and InflammaTION) in Persons With Multiple Sclerosis Study
Brief Title: the EXPOSITION Study
Acronym: EXPOSITION
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Pavia (Other)
Collaborators: National Research Council (Consiglio Nazionale delle Ricerche) (Unknown); IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 0040083/23
Record Dates: First submitted 2024-02-09; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Environmental Exposure; Lifestyle Factors
Keywords: multiple sclerosis; exposome; microRNA; cytokines; microbiome; neurofilament; air pollution; urbanization; lifestyle; nutrition; physical activity; inflammation
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Motor Activity; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with Multiple sclerosis: Age ≥ 18 years
  * Diagnosis of MS according to 2017 McDonald criteria
  * Relapsing-remitting (RR) MS
  * Residence in the provinces of Pavia or Milan (Italy)
  * Informed consent form signed

SUMMARY:
This is a cross-sectional study to evaluate the variation of biological biomarkers of oxidative stress and inflammation in response to the external exposome, in people with Multiple Sclerosis (pwMS).The objective is to study the variation of biological biomarkers of oxidative stress and inflammation in response to external exposome in pwMS, controlling for other biomarkers (cytokine, neurofilaments, microbiome), gender, age, anthropometric measurements, vitamin D levels and medical history. Specifically, the variation of microRNAs is defined as the primary outcome, in response to urban air pollution, urbanization, lifestyle and quality of life components of the external exposome. Following the functional exposome approach:(1)Information on a pwMS sample about socio-demographic characteristics and medical history will be collected and specific components of the (2) On the same pwMS sample, the internal exposome variation will be measured. MicroRNA levels and gut and nasal microbiota alpha- and beta-diversity and relative bacterial abundances will be considered as biomarkers of oxidative stress and inflammation. At the same time, cytokines and neurofilament proteins (NfL) will be measured as biomarkers of neurodegeneration and axonal damage. Adults (≥ 18 years) pwMS, with relapsing-remitting course, diagnosis of MS according to 2017 McDonald criteria and residing in Pavia or Milan (Italy) will be included. Potentially eligible pwMS will be screened by a neurologist expert in MS who will verify that all the inclusion criteria will be fulfilled. To validate variation among 7 selected MS diagnostic miRNA, in response to urban air pollution, urbanization, lifestyle and quality of life components of the external exposome, the differential expression (ΔCT) for each miRNA will be considered as the outcome measure. Two hundred eligible pwMS who meet the inclusion criteria and sign the informed consent will be included in the study, to consider 15% dropout at the blood sampling stage.

ELIGIBILITY:
Inclusion Criteria:

* We will include persons with Multiple Sclerosis (pwMS) attending the Centro Sclerosi Multipla of the IRCCS Fondazione C. Mondino of Pavia, according to the following inclusion criteria:

  * Age ≥ 18 years
  * Diagnosis of MS according to 2017 McDonald criteria
  * Relapsing-remitting course (RR)
  * Routine clinical examinations scheduled in the study period September 15, 2023, to March 15, 2024,
  * Residing in the provinces of Pavia and Milano
  * Informed consent form signed

Exclusion Criteria:

* Exclusion criteria will involve people refusing to participate in the study or people not completely meet the inclusion criteria. Potentially eligible pwMS will be screened by a neurologist expert in MS who will verify that all the inclusion criteria will be fulfilled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with Multiple Sclerosis (pwMS) attending the Centro Sclerosi Multipla of the IRCCS Fondazione C. Mondino of Pavia will be eligible, according to the following inclusion criteria:
  * Age ≥ 18 years
  * Diagnosis of MS according to 2017 McDonald criteria
  * Relapsing-remitting course (RR)
  * Routine clinical examinations scheduled in the study period September 15, 2023, to March 15, 2024,
  * Residing in the provinces of Pavia and Milano
  * Informed consent form signed
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
microRNAs | from March 2024 to July 2024 visit
  The differential expression of a set of 7 specific circulating plasma microRNAs from the blood of each pwMS will be measured. The set of miRNAs has been already selected based on their significant deregulated expression in MS, as evidenced in a bioinformatic analysis conducted using computational resources. A portion of serum samples will be collected and immediately frozen at -20°C. After being transported, serum samples will be thawed and the circulating RNAs will be extracted. After a step of microRNA specific reverse transcription, the copy-DNA obtained will be used as the template for Real Time-qPCR analyses of selected miRNAs by Singleplex TaqMan microRNA assay reactions.The method of Livak et al. will be applied for the comparative analysis of the relative expression of the selected microRNAs in serum samples, considering different combinations of the external exposome variables.
Air quality | from March 2023 to July 2023
  Spatial information on pollutants such as PM10, PM2.5, PM1.0 expressed in microg/m3, nanoparticulate (n/cm3), and black carbon (microg/m3) from CAMS and CHIMBO databases and from Sentinel-5P TROPOMI will be included as gridded emissions in 0.1° x 0.1° (long-lat) resolution for the whole time series (daily values), from March 2023 onwards from the Pavia and Milano provinces. Large Eddy Simulations will be carried out over such areas with a high spatial-temporal resolution for estimating - in a quantitative manner - the 3D pollutants concentration at the street level.The grid will be further subdivided into the municipalities of the two provinces and a "personal exposure" will be also assessed, based on the geographic position of each pwMS derived from the residence address (geo-positioning).
Nutritional assessment | from March 2024 to July 2024
  The dietary habits of the participants will be evaluated with the use of a validated food frequency questionnaire (FFQ) adapted to the Italian population and adjusted based on current food trends, such as the consumption of plant-based milk and meat. Detailed information about the daily food consumption of pwMS will be gained through a 24-h dietary recall.
Neurofilament (NfL) | from March 2024 to July 2024
  Human NfL will be assessed on plasma samples by Simple Plex assay (ProteinSimple, CA, USA) on Ella device (ProteinSimple, CA, USA), according to the manufacturer's instructions. Calibration of Ella will be performed using the incartridge factory standard curve, and plasma samples will be measured with a 1:2 dilution in Sample Diluent (ProteinSimple, CA, USA). A single well was used for each sample as triplicates assays are automatically performed in Simple Plex assay microfluidic platform. The LLOQ is 2.70 pg/ml; the upper limit of quantification is 10,290.00 pg/ml.
Cytokines | from March 2024 to July 2024
  Serum levels of IL1-beta, IL2, IL4, IL6, IL-10, IL12, IL17, IL22, IL23, TGF-beta, GM-CSF, TNF-alpha, IFN-gamma expressed in pg/mL will be assessed by using CXCL10 (performed using Simple Plex , R&D and commercial ELISA kit).
the Body Mass Index (BMI) | from March 2024 to July 2024
  Weight in kg and height in m will be measured in order to calculate the Body Mass Index (BMI) as the ratio of weight (kg) to height (m) squared.
Physical activity | from March 2024 to July 2024
  Physical activity levels will be evaluated by using the International Physical Activity Questionnaires (IPAQ) . The questionnaire is composed of 7 questions concerning the last 7 days levels of moderate, vigorous and sedentary physical activity. The metabolic equivalent of tasks (MET) will be calculated using the frequency and duration of physical activity and will be reported as MET-min/wk.
Quality of life related to MS | from March 2024 to July 2024
  Quality of life will be evaluated by Multiple Sclerosis Quality of Life-29 (MSQOL-29), a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument.
Sleep Quality | from March 2024 to July 2024
  Sleep quality will be measured by the Pittsburgh Sleep Quality Index (PSQI) questionnaire. The questionnaire consists of 9 multiple-choice items divided into 5 different components related to subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication and daytime dysfunction. The global PSQI score will be obtained by considering the scores of all the components and it ranges from 0 to 13. The PSQI cut-off of 5 or above indicates poor sleep quality.
Smoking habits | from March 2024 to July 2024
  Cigarette smoking habits will be registered considering patients who are smoking, never smoked and quit smoking. The number of cigarettes smoked per day and the years of smoking will be recorded for smokers. Ex-smokers will be asked the number of years not smoking, the number of years that have smoked and the number of cigarettes smoked per day during their smoking years.
Dietary supplements use | from March 2024 to July 2024
  Dietary supplements use will be assessed based on the type and nutrients included in the dietary supplements, their dose and their frequency of use.
Adherence to Mediterranean diet | from March 2024 to July 2024
  Adherence to the Mediterranean dietary model will be assessed by applying the MEDI-LITE score. The MEDI-LITE score is based on a questionnaire, which investigates the frequency of consumption of nine classes of food. The final score varies from 0 (low adherence) to 18 (high adherence). Overall, subjects who will obtain a score higher than 9 will have a significantly increased adherence to the Mediterranean Diet.
Effect of diet on inflammation | from March 2024 to July 2024
  The Dietary Inflammatory Index (DII) will be also calculated to quantify the overall effect of diet on inflammatory potential. The DII will be calculated based on the daily food consumption and then based on it the food parameters included in DII will be evaluated, such as vitamins, macronutrients, minerals, green/black tea and others.
waist and height ratio (WHtR) | from March 2024 to July 2024
  The waist circumference and (cm) height (cm) will be measured in order to calculate their ratio (WHtR), a good predictor of abdominal adiposity in adults, will be also calculated.
Bioelectrical impedance | from March 2024 to July 2024
  Bioelectrical impedance analysis will be used for the analysis of phase angle (PhA), which is considered an indicator of cellular health and malnutrition.

SECONDARY OUTCOMES:
Microbiome and biological biomarkers of oxidative stress and inflammation | from March 2024 to July 2024
  The percentage of each bacterial operational taxonomic units (OTUs) was investigated separately for each sample, providing relative abundance data among the samples based on the the relative numbers of reads within each.
  Microbial profiles will be evaluated in terms of
  1. Biodiversity (alpha-diversity), estimating the number of taxa in each sample and statistically comparing estimates across the experimental groups;
  2. Composition (beta-diversity), evaluating the pairwise similarity among the samples and clustering them according to their distances;
  3. Bacterial groups (relative abundances), evaluating whether a bacterial taxon is significantly increased or depleted in pwMS belonging to the different exposome variables under investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Tavazzi, Principal Investigator — Neurological Institute-Foundation IRCCS Casimiro Mondino, Pavia, Italy
Locations (1):
- IRCCS Foundation C. Mondino, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Monti MC, De Giuseppe R, Bertoli G, Alemayohu MA, Al-Naqeb G, Ballante E, Bergamaschi R, Camboni T, Ceccarani C, Ceriani C, Colombo E, Consolandi C, Costabile F, Decesari S, Gallivanone F, Galuzzi BG, Gastaldi M, Gervasoni C, Gugiatti S, Itri T, Kalmpourtzidou A, Landi TC, Lanzotti A, Dico AL, Loperfido F, Maccarini B, Mazza A, Montomoli C, Oddone E, Paulin N, Pellizzer C, Pernetti R, Scarabotto A, Sellaro F, Severgnini M, Summa D, Vivone G, Porro D, Cena H, Tavazzi E. Exposome, oxidative stress and inflammation in persons with multiple sclerosis: the EXPOSITION study protocol. Front Public Health. 2025 Oct 22;13:1688158. doi: 10.3389/fpubh.2025.1688158. eCollection 2025. PMID 41200026